CLINICAL TRIAL: NCT02539420
Title: A Prospective, Randomized Trial of Early Versus Delayed BiPAP Administration or Non-positive Pressure Therapy in the Management of Pediatric Status Asthmaticus
Brief Title: A Prospective Trial of BiPAP Administration vs. Non-positive Pressure Therapy for Pediatric Status Asthmaticus
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: Feinstein Institute for Medical Research (Other)
Responsible Party: Principal Investigator, Sandeep Gangadharan, Attending physician, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-245
Record Dates: First submitted 2015-08-26; First posted 2015-09-03 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: Status Asthmaticus
MeSH Terms: conditions — Status Asthmaticus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Patients assigned to the "control" group will receive any treatment for status asthmaticus that does not entail use of positive pressure ventilation.
- Late BiPAP treatment (Experimental): Patients assigned to the "late treatment" group will be started on BiPAP greater than 6 hours after randomization.
  Interventions: Device: BiPAP treatment
- Early BiPAP treatment (Experimental): Patients assigned to the "early treatment" group will be started on BiPAP as soon as possible after randomization.
  Interventions: Device: BiPAP treatment

INTERVENTIONS:
Device: BiPAP treatment — Patients will receive BiPAP (via Respironics V60 or Vision BIPAP device) as part of their treatment for status asthmaticus
  Arms: Early BiPAP treatment; Late BiPAP treatment

SUMMARY:
Though BiPAP is an increasingly common tool used by pediatric critical care physicians and there is promising data suggesting a role for BiPAP in the management of status asthmaticus, more information is needed to more definitively clarify the extent of its benefit, as well as when during an asthma exacerbation and in whom it is the most beneficial. In this study, which is among the first randomized studies of BiPAP use for status asthmaticus in the pediatric population, the investigators hope to better elucidate these issues to help guide clinicians' future management decisions.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of asthma exacerbation
* Admitted to Cohen Children's Medical Center (CCMC) PICU
* CCMC respiratory severity score of 6 or higher at the time of enrollment
* Prior history of asthma or reactive airway disease

Exclusion Criteria:

* No prior history of asthma or reactive airway disease
* Facial or airway anomalies precluding BiPAP mask use
* Tracheostomy
* Lack of airway protective reflexes
* Neurologic or musculoskeletal abnormalities affecting respiration
* Underlying cardiovascular problems that may be negatively affected by positive pressure ventilation
* Intracranial problems (such as in the setting of head injury) that may be negatively affected by positive pressure ventilation
* Respiratory compromise for which emergent endotracheal intubation or non-invasive positive pressure ventilation is warranted as determined by the on-service attending physician

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2016-04; Primary Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Clinical Asthma Scores | 3 hours after enrollment
  Both PRAM and CCMC clinical asthma scores

SECONDARY OUTCOMES:
Dyspnea Scores | 0 hours, 3 hours, 6 hours, 9 hours, 12 hours, 24 hours, and 36 hours after enrollment
  Modified Borg Scale and Wong Baker Faces Scale
BiPAP Tolerance | Hospitalization
  Tolerability of BiPAP will be determined by patients keeping the mask on and agreeing to remain on the machine for the intended treatment period.
Length of stay in intensive care unit (ICU) | ICU stay -- Expected to be approximately 3 days on average
Length of stay in hospital | Hospital length of stay -- Expected to be approximately 5 days on average
Side effects or adverse events | Hospitalization
Clinical Asthma Scores | 0 hours, 6 hours, 9 hours, 12 hours, 24 hours, and 36 hours after enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Gangadharan, MD, Principal Investigator — Cohen Children's Medical Center